CLINICAL TRIAL: NCT00222079
Title: Pilot Study to Evaluate Esomeprazole (Nexium) in Treating Gastro-esophageal Reflux in Patients With Head and Neck Cancer With Prior External Beam Radiation Therapy: a Randomized, Prospective, Placebo-controlled, Double-blind Study.
Brief Title: Evaluation of Esomeprazole in Treating Gastro-esophageal Reflux Disease (GERD) in Head and Neck Cancer Patients Exposed to Radiation Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Project canceled due to the implementation of IMRT, fewer patients reporting xerostomia.
Sponsor: Douglas Trask (Other)
Responsible Party: Sponsor-Investigator, Douglas Trask, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 200308067
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Gastro-esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole (Nexium)

SUMMARY:
The purpose of this research study is to measure acid reflux into the throat both before and after medical treatment in people who have had radiation therapy to their head and neck for the treatment of cancer. Many people who have received head and neck radiation therapy develop a dry mouth as a result of the radiation damage to their saliva glands. In addition to the discomfort associated with a dry mouth, the decrease in saliva may increase the severity of gastro-esophageal reflux disease (acid reflux). Acid reflux occurs when acid escapes from your stomach into your throat. You may not have any symptoms of acid reflux, but often it can cause symptoms of heartburn or chest discomfort.

Acid reflux can be treated once it is diagnosed. Treatment consists of dietary changes, behavioral alterations, and medication. Medications are available that decrease the amount of acid in your stomach. Diagnosis of acid reflux is made with a pH-probe to test for acid in your throat.

DETAILED DESCRIPTION:
The annual incidence of squamous cell carcinoma of the head and neck (SCCHN) is 40,000 cases per year in the US and 60,000 cases per year in Europe. Radiation therapy is employed in combination with chemotherapy in primary treatment or as adjuvant therapy for over half of patients with SSCHN.

A high incidence of pathologic laryngopharyngeal reflux and gastroesophageal reflux is observed in patients with head and neck cancer. When treatment for the cancer includes radiation therapy, an incidence of 90% has been reported [2]. Although the interplay between acid reflux and the development of head and neck cancer remains unclear, there is a strong argument that radiation therapy worsens the problem by muting the body's ability to neutralize acid.

Radiation therapy is extensively used in the treatment of squamous cell carcinoma of the head and neck. Radiation therapy works by exploiting a survival differential between malignant cells and normal cells. Simply stated, the malignant cells are more likely to die with radiation when compared to normal non-malignant cells. However, not all normal cells respond equally and some normal tissues have marked sensitivity to radiation damage. Salivary glands are one such radiosensitive tissue that is permanently destroyed with external-beam radiotherapy.

Damage to salivary tissues by radiation decreases their ability to excrete saliva. This is supported by Olmos et al, who used salivary scintigraphy on both irradiated and non-irradiated patients and found that 84% of those irradiated had total or partial disturbance in both baseline and stimulated function. Of those treated with greater than 4500cGy, salivary excretion was almost invariably impaired. Xerostomia is the term for the dry mouth, which can result from this loss.

In addition to the volume of the saliva, the contents of the saliva are also important. Helm et al. "…evaluated the properties of human saliva relevant to its potential contribution to esophageal acid clearance." By measuring the capacity for acid neutralization and plotting titration curves, they identified that saliva and especially its bicarbonate content play an important role in neutralization of esophageal acid in both resting and lozenge-stimulated states.

As saliva plays an active role in the neutralization of esophageal acid and its clearance from the esophagus, loss of saliva is predicted to increase the severity and incidence of reflux as the protective effect of saliva's ability to clear and neutralize acid reflux is diminished. Korsten et al., assessed the effects of chronic xerostomia on parameters of gastroesophageal reflux and esophagitis and reported markedly impaired clearance of acid from the esophagus and abnormal 24-hour intra-esophageal pH studies from a cohort of male patients with xerostomia.

Medications are available to increase salivary flow but these are often minimally effective and poorly tolerated. Decreasing stomach acid production is an alternative method of mitigating the effect of GERD in these patients.

Esomeprazole has been proven beneficial in the treatment of gastroesophageal reflux disease and is anticipated to be beneficial in treating SCCHN patients treated with external-beam radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. History of head and neck cancer
3. Radiation Therapy (external beam or IMRT)

   1. Must have received equal or greater than 5000 cGy cumulative dose
   2. Must have complaint of xerostomia
   3. Greater than three month interval since radiation treatment

Exclusion Criteria:

1. Subjects unable to tolerate pH-probe in past
2. Subjects currently on proton-pump inhibitor (PPI) or H-2 receptor antagonist therapy
3. Prior history of esophago-gastric surgery
4. Symptoms of gastrointestinal bleeding (melena, hematemesis)
5. Known hepatic cirrhosis or esophageal varices
6. Prior esophageal perforation
7. Pregnant, nursing or not likely to be using adequate contraceptive measures
8. Subjects not predicted to survive duration of study
9. Subjects with allergies or sensitivities to proton-pump inhibitors
10. Psychological, familial, sociological or geographical conditions which do not permit Study follow-up and compliance with study protocol
11. Subjects predicted to undergo surgery, chemotherapy or radiation therapy for head and neck cancer during the course of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-11 (Actual); Primary Completion 2007-10 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas K trask, MD. Ph.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Department of Otolaryngology, Iowa City, Iowa, United States